CLINICAL TRIAL: NCT03708770
Title: everlinQ Endovascular Access System Enhancements (EASE) Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: C. R. Bard (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CD-0015
Record Dates: First submitted 2018-07-26; First posted 2018-10-17 (Actual); Results first posted 2019-06-14 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: Chronic Kidney Diseases
MeSH Terms: conditions — Renal Insufficiency, Chronic

ARMS (1):
- endoAVF (Other)
  Interventions: Device: everlinQ endoAVF System

INTERVENTIONS:
Device: everlinQ endoAVF System

SUMMARY:
Prospective, single-center study to evaluate the everlinQ System when used to create an endoAVF in hemodialysis patients.

DETAILED DESCRIPTION:
A total of up to 50 subjects will be enrolled and will undergo an endoAVF creation procedure using the everlinQ System. All subjects will be followed for up to 12 months post index procedure based on Investigator's discretion.

ELIGIBILITY:
Inclusion Criteria:

1. Eligible for a native arteriovenous fistula.
2. Adult (age >18 years old).
3. Established, non-reversible kidney failure requiring hemodialysis (including pre-dialysis patients).
4. Target vein diameter(s) ≥ 2.0 mm or large enough to accommodate device diameter.
5. Target artery diameter ≥ 2.0 mm or large enough to accommodate device diameter.
6. Estimated life expectancy > 1 year.
7. Patient is free of clinically significant conditions or illness within 30 days prior to the AV fistula that may compromise the procedure

Exclusion Criteria:

1. Known central venous stenosis or central vein narrowing > 50% based on imaging on the same side as the planned AVF creation.
2. Upper extremity venous occlusion(s) and/or vessel abnormality(ies) on the same side as the planned AVF creation that precludes endovascular AVF creation by everlinQ System as deemed by the interventionalists' clinical judgment.
3. Prior surgically created access in the planned treatment location.
4. Functioning surgical access in the planned treatment arm.
5. Pregnant women.
6. New York Heart Association (NYHA) class III or IV heart failure.
7. Hypercoagulable state.
8. Known bleeding diathesis.
9. Immunosuppression, defined as use of immunosuppressive medications used to treat an active condition.
10. Documented history of drug abuse including intravenous drugs within six months of AVF creation.
11. "Planned" concomitant major surgical procedure within 6 months of enrollment or previous major surgery within 30 days of enrollment.
12. Currently being treated with another investigational device or drug.
13. Known allergy to contrast dye which cannot be adequately pre-medicated. CD-0015 Rev 02 - EASE Study Clinical Protocol CONFIDENTIAL Page 8 of 16
14. Known adverse effects to sedation and/or anesthesia which cannot be adequately pre-medicated.
15. Patients who do not have an ulnar or radial artery.
16. At the time of procedure distance between target artery and vein will not allow magnets to align vessels sufficiently to create the fistula.
17. Evidence of active infections on the day of the index procedure.
18. Written informed consent not obtained.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2015-07-27 (Actual); Primary Completion 2017-06-19 (Actual); Study Completion 2017-06-19 (Actual)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First subject enrolled July 27, 2015 and last subject enrolled November 8, 2016. Last subject follow-up was June 19, 2017.
Groups:
- endoAVF: everlinQ arteriovenous fistula (endoAVF) System
Period: Overall Study
Arm/Group | endoAVF
Started | 32
Completed | 22
Not Completed | 10

BASELINE CHARACTERISTICS:
Groups:
- endoAVF: everlinQ endoAVF System
Arm/Group | endoAVF
Number analyzed (Participants) | 32
Age, Customized [Mean (Standard Deviation); unit: Years]
  Age of Participants | 50.9 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 32
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Paraguay | 32
Fistula Type [Count of Participants; unit: Participants]
  Ulnar-Ulnar | 12
  Radial-Radial | 20
Access Arm [Count of Participants; unit: Participants]
  Right | 7
  Left | 25
Access Artery [Count of Participants; unit: Participants]
  Radial | 19
  Brachial | 9
  Ulnar | 4
Access Vein [Count of Participants; unit: Participants]
  Radial | 17
  Brachial | 13
  Ulnar | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Protocol-Defined endoAVF Maturation
Description: Protocol-defined endoAVF maturation is defined as endoAVF that is free of stenosis or thrombosis, with brachial artery flow at least 500ml/min and at least 4 mm vein diameter (as measured by duplex ultrasound) OR subject was dialized using 2 needles.
Time Frame: Through 6 months post-index procedure
Measure: Count of Participants; unit: Participants
Arm/Group | endoAVF
Number analyzed (Participants) | 32
Participants | 29

2. Primary Outcome: Number of Participants With Device-Related SAEs
Description: The safety Endpoint is protocol-defined as Device-Related SAE at 3 months.
Time Frame: 3 months following AVF creation
Measure: Count of Participants; unit: Participants
Arm/Group | endoAVF
Number analyzed (Participants) | 32
Participants | 0

3. Secondary Outcome: Number of Days to Fistula Maturation
Description: Defined as the number of days between the date of AVF creation and the date of endoAVF maturation (based on primary efficacy endpoint definition of maturation).
Time Frame: Days from Index Procedure
Measure: Mean (Standard Deviation); unit: Days from Index Procedure
Arm/Group | endoAVF
Number analyzed (Participants) | 32
Days from Index Procedure | 9.2 (19.1)

4. Secondary Outcome: Percentage of Participants With Secondary Patency at 6 Months Post-Index Procedure
Description: Time from endoAVF creation until access abandonment. Abandonment due to renal transplant receipt was not included in this endpoint assessment.
Time Frame: 6 months post-index procedure
Measure: Number; unit: Percentage of participants
Arm/Group | endoAVF
Number analyzed (Participants) | 32
Percentage of participants | 86.8
Statistical Analysis 1: Comparison: endoAVF; This was not a hypothesis-driven study. Therefore, there were no primary effectiveness or safety endpoints. The Secondary Patency endpoint was calculated using a Kaplan-Meier analysis; Test type: Other — No power calculation was performed for this study; The Secondary Patency rate was determined via Kaplan-Meier methods

5. Secondary Outcome: Primary Patency at 6 Months Post-index Procedure
Description: Primary Patency is defined as the interval following the index intervention until the next clinically driven reintervention at the original treatment site to maintain or reestablish patency or loss of endoAVF patency. The primary patency rate is determined via Kaplan-Meier methods and based on the time of endoAVF creation until any intervention designed to maintain or reestablish patnecy or endoAVF abandonment.
Time Frame: 6 months post-index procedure
Measure: Number; unit: Percentage of participants
Arm/Group | endoAVF
Number analyzed (Participants) | 32
Percentage of participants | 83.3
Statistical Analysis 1: Comparison: endoAVF; This was not a hypothesis-driven study. Therefore, there were no primary effectiveness or safety endpoints. The Primary Patency endpoint was calculated using a Kaplan-Meier analysis; Test type: Other — No power calculation was performed for this study; The primary patency rate was determined via Kaplan-Meier methods

6. Secondary Outcome: Number of Participants Per Catheter Exposure Type
Description: Number of participants with Central Venous Catheters (CVC), endoAVF only access, CVC + endoAVF access, and not reciving dialysis at 3 and 6 months post-index procedure.
Time Frame: 1-7 days, 30 days, 3, and 6 months post-index procedure
Population: Number of participants (n) for each follow-up period varies from total participants in the study (N=32) according to the number of participants that attend follow-up and/or had data relevant to the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | endoAVF
Number analyzed (Participants) | 32
Participants
  CVC only at 1-7 days post index procedure | 31
  EndoAVF only at 1-7 days post index procedure | 0
  CVC & endoAVF at 1-7 days post index procedure | 0
  No dialysis at 1-7 days post-index procedure | 1
  CVC only at 30 days post-index procedure: number analyzed (Participants) | 28
  CVC only at 30 days post-index procedure | 26
  EndoAVF only at 30 days post-index procedure: number analyzed (Participants) | 28
  EndoAVF only at 30 days post-index procedure | 1
  CVC & endoAVF at 30 days post-index procedure: number analyzed (Participants) | 28
  CVC & endoAVF at 30 days post-index procedure | 0
  No dialysis at 30 days post-index procedure: number analyzed (Participants) | 28
  No dialysis at 30 days post-index procedure | 1
  CVC only at 3 months post-index: number analyzed (Participants) | 16
  CVC only at 3 months post-index | 5
  EndoAVF only 3 months post-index: number analyzed (Participants) | 16
  EndoAVF only 3 months post-index | 10
  CVC + endoAVF at 3 months post-index: number analyzed (Participants) | 16
  CVC + endoAVF at 3 months post-index | 0
  No dialysis at 3 months post-index: number analyzed (Participants) | 16
  No dialysis at 3 months post-index | 1
  CVC only at 6 months post-index: number analyzed (Participants) | 26
  CVC only at 6 months post-index | 7
  EndoAVF only 6 months post-index: number analyzed (Participants) | 26
  EndoAVF only 6 months post-index | 19
  CVC + endoAVF at 6 months post-index: number analyzed (Participants) | 26
  CVC + endoAVF at 6 months post-index | 0
  No dialysis at 6 months post-index: number analyzed (Participants) | 26
  No dialysis at 6 months post-index | 0

7. Secondary Outcome: Number of Participants With Technical Success
Description: Technical success is defined as verification that an endoAVF has been created and remains patent 1-7 days after the index procedure. Patency is determined by experienced examiner as the presence of a bruit that is detected with stethoscope, or presence of thrill, or via Duplex Ultrasound, or via angiogram.
Time Frame: 1-7 days following index-procedure
Measure: Count of Participants; unit: Participants
Arm/Group | endoAVF
Number analyzed (Participants) | 32
Participants | 30

8. Secondary Outcome: Number of Endo-AVF-related Re-interventions
Description: The re-intervention rate for endo-AVF (defined as any intervention required to maintain or re-establish patency) was calculated at each available follow-up visit post-index procedure.
Time Frame: At 6 months follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | endoAVF
Number analyzed (Participants) | 32
Participants | 2

ADVERSE EVENTS:
Time Frame: Serious Adverse Events (SAEs) were collected through 6-months post-index procedure.
Description: Significant Adverse Events are defined as device or procedure-related adverse events (AE) that either, a) could be limb-threatening if not promptly identified or treated, or b) required additional therapy to reestablish patency of the endoAVF access circuit; irrespective of whether the event was an SAE. The SAE table combines both Significant Events and SAE events.
  Only AEs relevant to index-procedure, study device, access site or endoAVF were collected and are included in the Other AE table.
Arm/Group | endoAVF
All-Cause Mortality (participants affected / at risk) | 5/32
Serious Adverse Events (participants affected / at risk) | 2/32
Other Adverse Events (participants affected / at risk) | 7/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | endoAVF (N=32)
Bleeding/Hematoma (Blood and lymphatic system disorders) | 1 (1) — Procedure related.
Heart problems (Cardiac disorders) | 1 (1) — Not device or procedure-related.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | endoAVF (N=32)
Occlusion/Thrombosis (Vascular disorders) | 4 (4)
Occlusion/Stenosis (Vascular disorders) | 1 (1)
Bleeding/Hematoma (Blood and lymphatic system disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-07-05): https://cdn.clinicaltrials.gov/large-docs/70/NCT03708770/Prot_SAP_000.pdf